CLINICAL TRIAL: NCT00001254
Title: Evaluation of the Gastrinoma in Patients With Zollinger-Ellison Syndrome
Brief Title: Evaluating Pancreatic Tumors in Patients With Zollinger-Ellison Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 900137; 90-DK-0137
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-06-11

CONDITIONS: Zollinger Ellison Syndrome
Keywords: Zollinger-Ellison Syndrome; Natural History
MeSH Terms: conditions — Zollinger-Ellison Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients will Zollinger-Ellison Syndrome

SUMMARY:
This protocol concerns the approach to the localization, diagnosis of MEN1 and management of the tumor and the tissue samples in patients with Zollinger-Ellison syndrome. It details the diagnostic imaging tests to be used to localize the tumor, investigations for MEN1 the subsequent management of the tumor and tissue samples for research.

DETAILED DESCRIPTION:
This protocol concerns the approach to the localization and management of the tumor in patients with Zollinger-Ellison syndrome. It details the diagnostic imaging tests to be used to localize the tumor and the subsequent management of the tumor.

ELIGIBILITY:
* INCLUSION CRITERIA:

New patients will be evaluated initially as described in the protocol entitled, "Diagnostic evaluation of patients with suspected abnormalities of gastric secretion" (89-DK-0005).

Only those patients that are being treated under the protocol entitled, "Medical Therapy of Zollinger-Ellison Syndrome" (protocol # 89-DK-0015) will be entered into this tumor localization and management protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient population enrolled in protocol 89-DK-0015
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 1991-10-29 (Actual)

PRIMARY OUTCOMES:
To determine an approach to the localization and management of tumor in patients with ZES. | Yearly
  localization of tumor

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Jensen, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wolfe MM, Jensen RT. Zollinger-Ellison syndrome. Current concepts in diagnosis and management. N Engl J Med. 1987 Nov 5;317(19):1200-9. doi: 10.1056/NEJM198711053171907. PMID 3309661
- [Background] Andersen DK. Current diagnosis and management of Zollinger-Ellison syndrome. Ann Surg. 1989 Dec;210(6):685-703. doi: 10.1097/00000658-198912000-00001. PMID 2686566
- [Background] Creutzfeldt W, Arnold R, Creutzfeldt C, Track NS. Pathomorphologic, biochemical, and diagnostic aspects of gastrinomas (Zollinger-Ellison syndrome). Hum Pathol. 1975 Jan;6(1):47-76. doi: 10.1016/s0046-8177(75)80109-2. PMID 45919
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1990-DK-0137.html